CLINICAL TRIAL: NCT01090583
Title: Can Non-invasive Sampling Determine the Inflammatory Status of the Intra-uterine Environment?
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Daniel Kiefer, Fellow, Winthrop University Hospital
Other Study IDs: 09042
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Pregnancy
Keywords: Cytokines; Pregnancy; Cesarean
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: observational study, no specimens required.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cesarean Delivery Patients
  Interventions: Other: Specimen Collection

INTERVENTIONS:
Other: Specimen Collection — We will compare mediators from non-invasive samples (blood, urine, saliva, vaginal or cervical secretions) with traditional gold-standard invasive samples (amniotic fluid and placenta samples).

SUMMARY:
Preterm birth (birth before 37 weeks gestation) is a large problem in the United States and is a major cause of neonatal morbidity and mortality and childhood neurological disability. Despite significant advances in the care of pregnant mothers, the incidence of preterm labor is on the rise. There is growing recognition that cytokines and inflammatory mediators present at amniotic fluid and placenta play a fundamental role in regulating labor.

Cytokines are chemicals in the fluid that tell the body's immune system what to do. These (and other biomarkers) can be measured with a small amount (a few drops) of amniotic fluid. The researchers have previously shown that people at risk for preterm labor have higher cytokine levels. However, understanding the in-utero environment currently requires invasive sampling, such as amniocentesis, to determine cytokine concentrations. This procedure has inherent risks, causes patient discomfort and anxiety, and thus does not avail itself to routine use or repeated sampling, especially in non-high risk patients. Therefore, the researchers are looking for non-invasive sampling that can predict the in-utero environment.

To date, no studies have simultaneously evaluated different maternal-fetal compartments to determine the relationship of these markers among the compartments. Therefore, the purpose of this pilot study is to determine the differential expression of inflammatory mediators in various maternal-fetal compartments; specifically, vaginal fluid, cervical secretions, placenta, cord blood (arterial and venous), amniotic fluid, maternal serum, maternal urine, and maternal saliva.

The researchers seek to obtain fluid samples from nine maternal-fetal compartments and determine the inflammatory mediator expression in each. The timing of collection, location, and proposed studies for each of the samples is outlined in Table 1. In this pilot study, we plan to enroll 20 patients undergoing cesarean delivery.

After consent, the samples will be collected and given a unique Study ID number. No protected health information will be collected. In addition, there will be no link between the Study ID and patient identifiers. Therefore, we are not seeking HIPAA authorization at the time of consent. While none of these samples would routinely be collected as part of the standard of care, the collection procedures meet the criteria for minimal risk.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cesarean delivery
* Able to provide informed consent, including permission of storage of specimens
* No apparent major fetal abnormality

Exclusion Criteria:

* Major Fetal Malformation
* Rupture of membranes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The researchers seek to obtain fluid samples from nine maternal-fetal compartments and determine the inflammatory mediator expression in each. These mediators include cytokines, chemokines, and growth factors via the Bio-Plex™ Suspension Array system. In this study, we plan to enroll 20 patients undergoing cesarean delivery at term.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Cytokine Correlation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nazeeh Hanna, MD, Principal Investigator — Winthrop University Hospital